CLINICAL TRIAL: NCT02973685
Title: The Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy Compared With Transarterial Chemoembolization as Initial Treatment in Patients With Large Hepatocellular Carcinoma Staged BCLC A/B.
Brief Title: HAIC Versus TACE for Large Hepatocellular Carcinoma Staged BCLC A/B.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou No.12 People's Hospital (Other Government); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S023
Record Dates: First submitted 2016-11-20; First posted 2016-11-25 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: HepatoCellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Transarterial Chemoembolization; BCLC A/B
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; Pharmaceutical Preparations; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatic arterial infusion chemotherapy (Experimental): Procedure/Surgery: Hepatic arterial infusion chemotherapy Drug: Folfox Protocol. Hepatic intra-arterial infusion via the tumor feeding arteries of Oxaliplatin , fluorouracil, and leucovorin
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Folfox Protocol
- Transarterial chemoembolization (Active Comparator): Procedure/Surgery: Transarterial chemoembolization Drug: TACE Drug Protocol. Hepatic intra-arterial infusion with lipiodol mixed with chemotherapy drugs (EADM, lobaplatin, with or without MMC), and embolization with polyvinyl alcohol particles (PVA).
  Interventions: Procedure: Transarterial chemoembolization; Drug: TACE Drug Protocol

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — A standard hepatic artery catheter was introduced via the femoral artery percutaneously. Selective catheterization of the proper hepatic artery was performed using standard diagnostic catheters and fluoroscopic guidance. In the event of multiple arterial supply(including superior-mesenteric artery), the proportion of the liver supplied by each artery was estimated by the arteriogram. After optimal positioning of the catheter in dominant supplying artery to ensure minimal reflux, the catheter was fixed and connected with infusion tube. In the condition of multiple tumors on both left and right lobe, the gastroduodenal artery was embolized and the catheter was positioned in the hepatic proper artery for infusion. Folfox Protocol were infused through the fixed catheter sequentially.
  Arms: Hepatic arterial infusion chemotherapy
Procedure: Transarterial chemoembolization — Previous procedure was same with hepatic arterial infusion chemotherapy. After optimal positioning of the catheter, TACE Drug Protocol were injected.
  Arms: Transarterial chemoembolization
Drug: Folfox Protocol — oxaliplatin,leucovorin and 5-FU
  Other Names: Folfox for TAI
  Arms: Hepatic arterial infusion chemotherapy
Drug: TACE Drug Protocol — lipiodol mixed with chemotherapy drugs(EADM , lobaplatin, with or without MMC) followed by polyvinyl alcohol particles (PVA)
  Other Names: Drugs for transarterial chemotherapy and embolization
  Arms: Transarterial chemoembolization

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) compared with transarterial chemoembolization (TACE) in patients with large hepatocellular carcinoma staged BCLC A/B.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is the most widely used palliative treatment for hepatocellular carcinoma (HCC) patients. While a number of studies demonstrate poor effect of TACE for patients with large hepatocellular carcinoma staged BCLC A/B especially for those with tumor larger than 10 cm. Our previous prospective study also revealed similar results of large HCC patients treated with TACE. Recently, the results of our preliminary pilot study suggested that, compared with TACE, hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for HCC with large HCC. Thus, the investigators carried out this prospective randomized control to demonstrate the superiority of HAIC over TACE.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18-75 years;
* KPS≥70;
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL), simultaneously staged as BCLC A or BCLC B based on Barcelona Clinic Liver Cancer staging system.
* Patients must have at least one tumor lesion that can be accurately measured;
* The sum of diameters of all lesions longer than 10 cm with the maximum lesion longer than 7 cm.
* Diagnosed as unresectable with consensus by the panel of liver surgery experts;
* Re commanded treated by TAI or TACE with consensus by the panel of liver MDT;
* No past history of TACE, TAI, chemotherapy or molecule-targeted treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL;(b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits;(h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* Poor compliance that can not comply with the course of treatment and follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | 24 months

SECONDARY OUTCOMES:
Time to progression | 24 months
Adverse Events | 30 Days after HAIC
  Postoperative adverse events were graded based on CTCAE v4.03
Number of of Patients developed Adverse Events | 30 Days after HAIC
  Number of of patients who developed adverse event. Postoperative adverse events were graded based on CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (3):
- China (3):
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People's Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han X, Peng C, Ruan SM, Li L, He M, Shi M, Huang B, Luo Y, Liu J, Wen H, Wang W, Zhou J, Lu M, Chen X, Zou R, Liu Z. A Contrast-Enhanced Ultrasound Cine-Based Deep Learning Model for Predicting the Response of Advanced Hepatocellular Carcinoma to Hepatic Arterial Infusion Chemotherapy Combined With Systemic Therapies. Cancer Sci. 2025 Jul;116(7):1930-1940. doi: 10.1111/cas.70089. Epub 2025 Apr 29. PMID 40302359
- [Derived] Li QJ, He MK, Chen HW, Fang WQ, Zhou YM, Xu L, Wei W, Zhang YJ, Guo Y, Guo RP, Chen MS, Shi M. Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin Versus Transarterial Chemoembolization for Large Hepatocellular Carcinoma: A Randomized Phase III Trial. J Clin Oncol. 2022 Jan 10;40(2):150-160. doi: 10.1200/JCO.21.00608. Epub 2021 Oct 14. PMID 34648352
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/34648352